CLINICAL TRIAL: NCT06046885
Title: Effect of a Neuromuscular Electrostimulation Protocol on the Triceps Surae in Older Adults
Brief Title: Electrical Stimulation in Older Adults
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Gran Rosario (Other)
Responsible Party: Principal Investigator, Ivan Roulet, PT, University of Gran Rosario
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1820
Record Dates: First submitted 2023-06-27; First posted 2023-09-21 (Actual); Last update posted 2023-09-21 (Actual); Status verified 2023-06

CONDITIONS: Aged

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Electricalstimulation (Experimental)
  Interventions: Device: Neuromuscular electrical stimulation

INTERVENTIONS:
Device: Neuromuscular electrical stimulation — As regards the electrodes position, one proximal electrode on the gastrocnemius, which will be located below the popliteal fossa (at least 5cm below it) for a better position on the muscle belly; and one distal electrode, located at least 10 cm from the calcaneus.
  This protocol will last 20 minutes per session. The placement of the electrodes is as mentioned above, and the parameters to be used will be the following: a stimulation frequency between 35 and 80Hz, a pulse width between 150 and 200 µs, the intensity will be established individually using an intensity that generate a visible contraction of maximum intensity without generating pain. The duration of the contraction will be of 6 seconds with 30 seconds of rest.

SUMMARY:
Within the problems associated with population aging and its morbidities, the musculoskeletal system is involved in detrimental changes, compromising, in many cases, the functional capacity of the patient and their correct performance in the activities of daily living. Gait and stability are central axes to analyze and enhance in the elderly patient. Strategies for magnify these qualities are innumerable, although active exercise and electrostimulation comprise the most scientifically developed. Therefore, the objective of this study is to evaluate the effects of an electrostimulation (EE) program applied to the triceps surae in older adults on the temporo-spatial parameters of gait, stability and function.

DETAILED DESCRIPTION:
This is a quasi-experimental study with a sample of 13 volunteers. Patients of both genders and over 60 years old will be potential candidates for participating in the study. Volunteers will be invited to participate in the study through social networks and e-mail.

The study will be conducted in 12 experimental sessions on different days and 2 assessment days. During assessment sessions several measurements will be performed, including: balance (will be assessed using a balance tracking system balance plate) function (will be assessed by using the Short Physical Performance Battery) and gait (will be assessed using the Legsys device employing a 4 meter walk test).

The G-Power program (version 3.1.5, Franz Faul, Universität Kiel, Kiel, Germany) was used to perform the one-tailed sample calculation using a previous study . The isometric strenght of gastrocnemius was chosen as the main variable with an effect size of 0.70. The alpha level was set at 5%, and the estimated sampling power was 80%. The software returned a total sample of 13 individuals.

ELIGIBILITY:
Inclusion Criteria:

. To have signed the informed consent.

Exclusion Criteria:

* Surgical history of the lower extremities
* Uncontrolled neurological, metabolic disease
* Uncontrolled cardiac disease
* Uncontrolled respiratory disease

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2023-06-20 (Actual); Primary Completion 2024-08-20 (Estimated); Study Completion 2024-11-20 (Estimated)

PRIMARY OUTCOMES:
Change in ankle plantar-flexion strength | At baseline and 6 weeks later
  The ankle plantar-flexion strength will be measured with a wii balance board with the subject seated. A strap was placed distally on the thigh and passed directly over the external malleolus. The subject was asked to pull against the strap by extending his ankle while pushing with the sole of their foot and trying to lift the heel.

SECONDARY OUTCOMES:
Function | At baseline and 6 weeks later
  The function was assessed by using the Short Physical Performance Battery. This is a series of 3 tests to assess lower extremity physical function: a 4-meter walk at usual pace, time to complete 5 unassisted chair stands, and 3 standing balance tests. The scores range from 0 (worst performance) to 12 (best performance).
Function | At baseline and 6 weeks later
  Function was assessed using the Timed Up and Go test, this test uses the time (in seconds) that a person takes to rise from a chair, walk three meters, turn around 180 degrees, walk back to the chair and sit down while turning 180 degrees.
Change in balance | At baseline and 6 weeks later
  Balance will be assessed using a balance tracking system balance plate (Balance Tracking Systems, San Diego, CA). Participants stood on the plate for six testing trials. The first three measurement were made with bipedal stance and eyes closed, for about 30 seconds. The next three assessments were made with monopodal support on the right foot and the las 3 measurements were made with monopodal support on the left foot each monopodal repetition last 15 seconds.
Change in handgrip strength | At baseline and 6 weeks later
  The handgrip was assessed using a Jamar dynamometer while the subjects were sited.
Change in gait speed | At baseline and 6 weeks later
  The gait speed was assessed by using the time that a person takes to walk 4 meters distance. The test also included an acceleration phase of 2,5 meters, and a deceleration phase of 2,5 meters too.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Gran Rosario, Rosario, Santa Fe Province, Argentina